CLINICAL TRIAL: NCT00013026
Title: Trial of a Tailored Message Program to Implement CHF Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CPI 99-124
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Heart Failure
Keywords: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: CHF Self-management Education (Web-based Education)

INTERVENTIONS:
Behavioral: CHF Self-management Education (Web-based Education)

SUMMARY:
Congestive heart failure is a serious health problem in the United States and is associated with excessive morbidity and mortality. Several classes of medications have been shown to improve mortality in patients with CHF. Despite this these medications are widely under prescribed. Guidelines have been shown to improve patient outcomes and several guidelines on the management of CHF have been published. Implementation of guidelines is challenging and most strategies have focused on changing physician behavior. Patient-based interventions have been shown to be effective in implementing guidelines on CHF but they have been very labor intensive. A computer based intervention to implement CHF guidelines, if effective, would be beneficial.

DETAILED DESCRIPTION:
Background:

Congestive heart failure is a serious health problem in the United States and is associated with excessive morbidity and mortality. Several classes of medications have been shown to improve mortality in patients with CHF. Despite this these medications are widely under prescribed. Guidelines have been shown to improve patient outcomes and several guidelines on the management of CHF have been published. Implementation of guidelines is challenging and most strategies have focused on changing physician behavior. Patient-based interventions have been shown to be effective in implementing guidelines on CHF but they have been very labor intensive. A computer based intervention to implement CHF guidelines, if effective, would be beneficial.

Objectives:

Patients with CHF consume a significant proportion of healthcare resources, with exacerbations of CHF being the second most common reason for medical admission to VA medical centers. Therefore, the main objective is to understand the impact of a tailored education message program designed for direct use by patients on medical resource use. Other objectives include understanding the tools impact on patient compliance and quality of life.

Methods:

Patients have been randomized to one of two groups: 1) intervention group or the 2) control group. The intervention group receives the tailored education messages program. This program assesses patients� beliefs about compliance with medications, diet, and self-monitoring. Based on identified barriers to compliance, intervention patients receive a tailored educational message to dispel these beliefs and improve compliance. The control group interacts with a generic healthcare website. Patients in both groups are monitored for hospitalization; emergent care visits, compliance with prescribed treatment and quality of life

Status:

Project work is ongoing.

ELIGIBILITY:
Inclusion Criteria:

EF <40%, getting majority care at the VA, not enrolled in another CHF study, ability to read English.

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrence M. Shaneyfelt, MPH MD, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL; Catarina I. Kiefe, PhD MD, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (1):
- Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama, United States